CLINICAL TRIAL: NCT01950429
Title: Evaluation of Sickle Cell Liver Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130196; 13-DK-0196
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Sickle Cell Disease
Keywords: Microbiome; Sickle Cell Disease; Bone Marrow Transplant; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

- Sickle cell disease changes the shape of red cells. This makes them more likely to break down as they get stuck in small blood vessels. This leads to low red cell count and also damage to small blood vessels that supply many organs. One of the affected organs is the liver. Sickle cell disease and its treatment through blood transfusion can lead to significant liver damage. This disease also can cause the liver to regrow abnormally after damage. This can cause high blood pressure in the liver. Researchers want to know if curing sickle cell disease with a stem cell transplant improves liver damage.

Objectives:

- To explore specific factors that improve or worsen sickle cell liver disease after a stem cell transplant.

Eligibility:

- Adults ages 18 and older with sickle cell liver disease.

Design:

* Participation will take approximately 7 days over 2 years.
* Visit 1: participants will be screened with medical history and review of current treatment regimen.
* Visit 2: participants will return to the clinic for explanation of the study and physical exam. They will also have blood and urine tests, and scans of the liver.
* All participants will have a 2-night stay at the clinic. They will have a liver biopsy and a test of liver pressure. They will be sedated and a tube will be inserted in a vein in their neck.
* Participants who have a stem cell transplant will have a second biopsy about 24 months later.
* Over the 2-year study period, participants will have blood drawn 2-4 times and stool samples collected 2 times.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) causes multi-organ dysfunction and early death in affected individuals. Many succumb to complications of chronic organ dysfunction and eventual organ failure one of which is the liver.

Spectrum of sickle cell liver disease ranges from hepatic sequestration crisis, intrahepatic cholestasis, gallstones, non-cirrhotic portal hypertension, chronic sickle hepatopathy and cirrhosis to complications of the treatment of the disease including secondary iron overload and viral hepatitis. Though liver transplantation has been performed for SC-induced liver failure, a crude mortality rate of 60% makes it a poor choice. It is therefore imperative to identify patients with liver dysfunction and damage for possible early intervention.

Stem cell transplant is currently the only cure for SCD and at the NIH SCD hepatopathy is one of the indications for transplant. It is currently not known if stem cell transplant reverses SCD liver disease hence we intend to study and compare the nature of SCD liver disease pre and post stem cell transplant and in transplant ineligible patients. All SCD patients will be screened for liver disease prior to enrollment including fibroscan evaluation. Primary end point is histological evidence of regression of liver disease. Hence all patients in the transplant eligible arm will undergo liver biopsy pre and 12-24 months post transplant. Transplant ineligible patients will be offered liver biopsy when clinically indicated. Patients that have already undergone transplant will be included and their data evaluated retrospectively. Serum and plasma, liver tissue and stool samples will be evaluated extensively for parameters such as liver function tests, iron metabolism, clotting factors, and inflammatory markers including microbial products. The intention of the study is to use sickle cell disease as a model of predicting markers of progression and regression of liver disease.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. All age greater than 18 able to consent, male or female
  2. Capacity to provide written informed consent
  3. All ethnicities
  4. Sickle cell genotypes; Homozygous Hemoglobin S Disease, Heterozygous Hemoglobin SC and S beta thalassemia including SB+ and SB0
  5. Evidence of SCD liver dysfunction by abnormal liver laboratory parameters in at least 2 of the following; alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), direct and total serum bilirubin > 1 times ULN)

EXCLUSION CRITERIA:

1. If not taking measures to prevent pregnancy during the period of study
2. Incapacity to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sickle cell disease (SCD) causes multi-organ dysfunction and early death in affected individuals (1-4). Many succumb to complications of chronic organ dysfunction and eventual organ failure one of which is the liver. Spectrum of sickle cell liver disease ranges from hepatic sequestration crisis, intrahepatic cholestasis, gallstones, non-cirrhotic portal hypertension, chronic sickle hepatopathy and cirrhosis to complications of the treatment of the disease including secondary iron overload and viral hepatitis. Though liver transplantation has been performed for SC-induced liver failure, a crude mortality rate of 60% makes it a poor choice (5). It is therefore imperative to identify patients with liver dysfunction and damage for possible early intervention.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Histological evidence of regression of liver disease in stem cell transplanted sickle cell patients measured by degree of improvement in Deugnier's and HAI score | 5 years
  To assess severity, rule out portal hypertension, judge prognosis and to help in decisions on altering management

SECONDARY OUTCOMES:
Clinical evidence of regression of liver disease in transplanted sickle cell patients. Evaluate relationship between change in liver disease, bile acids, microbiome and prevalence of infection in SCD. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All collected IPD.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and any additional supporting information will become available 6 months after publication.
Access Criteria: Any secondary use requests will be reviewed and approved by the PI Theo Heller, MD.

REFERENCES:
- [Background] Panepinto JA, Walters MC, Carreras J, Marsh J, Bredeson CN, Gale RP, Hale GA, Horan J, Hows JM, Klein JP, Pasquini R, Roberts I, Sullivan K, Eapen M, Ferster A; Non-Malignant Marrow Disorders Working Committee, Center for International Blood and Marrow Transplant Research. Matched-related donor transplantation for sickle cell disease: report from the Center for International Blood and Transplant Research. Br J Haematol. 2007 Jun;137(5):479-85. doi: 10.1111/j.1365-2141.2007.06592.x. Epub 2007 Apr 24. PMID 17459050
- [Background] Berthaut I, Guignedoux G, Kirsch-Noir F, de Larouziere V, Ravel C, Bachir D, Galacteros F, Ancel PY, Kunstmann JM, Levy L, Jouannet P, Girot R, Mandelbaum J. Influence of sickle cell disease and treatment with hydroxyurea on sperm parameters and fertility of human males. Haematologica. 2008 Jul;93(7):988-93. doi: 10.3324/haematol.11515. Epub 2008 May 27. PMID 18508803
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0196.html